CLINICAL TRIAL: NCT02656914
Title: Phase III, National, Multicenter, Randomized, Double-blind Clinical Trial to Evaluate the Efficacy and Safety of Irlanda-2 Association on the Treatment of Common Cold
Brief Title: Efficacy and Safety of Irlanda-2 Association on the Treatment of Common Cold
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMS1115
Record Dates: First submitted 2016-01-12; First posted 2016-01-15 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irlanda-2-Association (Experimental): Take 10 mL every 12 hours (2x/day), oral route.
  Interventions: Drug: Irlanda-2-Association
- Placebo (Placebo Comparator): Take 10 mL every 12 hours (2x/day), oral route.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Irlanda-2-Association — Take 10 mL every 12 hours (2x/day), oral route.
  Arms: Irlanda-2-Association
Drug: Placebo — Take 10 mL every 12 hours (2x/day), oral route.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy of the drug associations in the treatment of common cold

DETAILED DESCRIPTION:
Double blind,randomized, multicenter; Maximal experiment duration: 7 days; 03 visits; Safety and efficacy evaluation

ELIGIBILITY:
Inclusion Criteria:

* Participant within 48 hours of the onset of common cold symptoms: headache, sneezing, sore throat, nasal obstruction, cough, coryza and body pain;
* Signed consent.

Exclusion Criteria:

* Patients with any clinically significant disease that, in the investigator opinion, can´t participate in the study;
* Patients with any laboratory finding or image finding that, in the investigator opinion, can´t participate in the clinical trial;
* Patients with history of hypersensitivity to any of the formula compounds;
* Participation in clinical trial in the year prior to this study;
* Patients with vaccine reaction;
* Patients who have uncontrolled asthma. However, participants in use of pulmonary corticosteroids (alone or in combination with other products) will be allowed if they are in stable dose and diagnosed with controlled asthma;
* Patients with gastroesophageal reflux, gastric or duodenal ulcer or other serious disease of the gastrointestinal tract;
* Patients with diabetes mellitus type I and II;
* Pregnancy or risk of pregnancy and lactating patients;
* Patients in use of drugs that can interfere with flu symptoms evaluation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Determine efficacy of Irlanda-2-Association in the treatment of common cold symptoms. | 7 days

SECONDARY OUTCOMES:
Safety will be evaluated by the adverse events occurrences | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Allergisa, Campinas, São Paulo, Brazil